CLINICAL TRIAL: NCT01548352
Title: BAsel Syncope EvaLuation (BASEL IX) Study
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: BASEL IX
Record Dates: First submitted 2012-03-05; First posted 2012-03-08 (Estimated); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Syncope
Keywords: Syncope; Unconsciousness; Syncope, vasovagal, neurally-mediated; Syncope, cardiogenic; Cardiac arrhythmia; Sudden cardiac death; Syncopal episode
MeSH Terms: conditions — Syncope; Unconsciousness; Syncope, Vasovagal; Arrhythmias, Cardiac; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — EDTA Plasma; Heparin; Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
Syncope is a major health problem. In the emergency department (ED), the management of patients with syncope still remains a clinical challenge because underlying diseases and prognosis can be extremely various. Structural heart disease and primary electrical disorders are major risk factors for sudden cardiac death and mortality in patients with syncope. In contrast, patients with reflex syncope and exclusion of structural heart disease have an excellent prognosis.

Therefore The investigators test the hypothesis that the use of a meticulous patient history, clinical examination and novel biomarkers can improve the rapid and accurate diagnosis of cardiac syncope in patients presenting to the ED and is able to improve risk stratification regarding adverse outcomes.

The prospective multicenter cohort study is designed to enroll 720 patients presenting with transient loss of consciousness within the last 12 hours to the ED. Blood samples for the measurement of novel biomarkers will be obtained at presentation.

All patients will be contacted by phone at 6, 12 and 24 months to determine major adverse events (death, resuscitation, recurrence of syncope, hospitalization for syncope).

DETAILED DESCRIPTION:
Background: Management of patients with syncope is a serious problem concerning 1-2% of emergency department (ED) visits. In 6-20% of these, syncope will be due to a cardiac origin. The rapid and accurate identification of these patients is an important unmet clinical need.

Aim: The aim of the study is to evaluate the diagnostic value of patient's history, clinical judgement and novel biomarkers, alone or in combination, in the diagnosis and risk stratification of patients > 40 years of age presenting with syncope to the ED.

Patients and Methods: This prospective, observational, international multicenter study is initially designed to enroll 720 adult patients > 40 years presenting to the ED with syncope within the last twelve hours. Patient history will be standardized using a predefined form. Treating physicians will be asked to quantify their clinical judgment regarding the presence of cardiac syncope. Digital 12-lead ECG will be recorded at presentation and stored electronically. Blood samples for the measurement of novel cardiovascular biomarkers (including copeptin, pro-endothelin-1, pro-adrenomedullin, natriuretic peptides and high-sensitive cardiac troponins) will be obtained at presentation and stored anonymized. Patients will be contacted by phone at 6, 12 and 24 months to determine major adverse events (death, resuscitation, recurrence of syncope, hospitalization for syncope) and results of follow-up examinations. The final diagnosis will be adjudicated by two independent experts after review of all documents pertaining to the individual patient after 6 months. The primary endpoint is to assess the performance of a standardized form of patient's history, clinical judgment and biomarkers, alone and in combination, in the diagnosis of a cardiac syncope, as adjudicated by two independent experts. Secondary endpoints include the accuracy of the above cited items in prognostic stratification and the determination of the cost-effectiveness of the best approach.

Clinical significance: A more accurate and more rapid diagnosis and risk stratification of cardiac syncope can significantly improve patient management and therefore reduce patient morbidity and treatment cost. Overall, we expect this study to provide novel insights, holding important scientific, clinical and economic implications.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the emergency department
* Age > 40 years
* Syncope within the last 12 hours
* Written informed consent

Exclusion Criteria:

* Age < 40 years
* Patients without loss of consciousness and with certain neurological causes (e.g. recurrent epilepsy, hemiplegia at presentation)
* No written informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the emergency department with syncope within the last 12 hours.
Sampling Method: Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2010-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic and prognostic value of various novel and established biomarkers, clinical assessment and detailed patient history | within 24 months
  To test the diagnostic performance of predefined elements of a standardized patient history, overall clinical judgement using a visual analogue scale, and novel biomarkers in the diagnosis of cardiac syncope in patients presenting to the ED.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Mueller, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (15):
- Baylor College of Medicine, Houston, Texas, United States
- Instituto Cardiovascular de Buenos Aires, Buenos Aires, Argentina
- Royal Brisbane and Women's hospital, Brisbane, Australia
- Klinikum Nürnberg, Nuremberg, Bavaria, Germany
- Sant'Andrea Hospital, Rome, Italy
- Christchurch Hospital, Christchurch, New Zealand
- Medical University of Silesia, Zabrze, Poland
- Spain (3):
  - Hospital del Mar, Barcelona
  - Hospital Clinic of Barcelona, Barcelona
  - Hospital Universitario Clínico San Carlos, Madrid
- Switzerland (5):
  - Kantonsspital Baselland, Liestal, Basel-Landschaft
  - Spital Lachen, Lachen, Canton of Schwyz
  - University Hospital Basel, Basel
  - Luzern Kantonsspital, Lucerne
  - University Hospital Zurich, Zurich

REFERENCES:
- [Derived] Zimmermann T, du Fay de Lavallaz J, Walter JE, Strebel I, Nestelberger T, Joray L, Badertscher P, Flores D, Widmer V, Geigy N, Miro O, Salgado E, Christ M, Cullen L, Than M, Martin-Sanchez FJ, Di Somma S, Peacock WF, Keller D, Costabel JP, Wussler DN, Kawecki D, Lohrmann J, Gualandro DM, Kuehne M, Reichlin T, Sun B, Mueller C; BASEL IX and SRS Investigators. Development of an electrocardiogram-based risk calculator for a cardiac cause of syncope. Heart. 2021 Nov;107(22):1796-1804. doi: 10.1136/heartjnl-2020-318430. Epub 2021 Jan 27. PMID 33504514
- [Derived] Zimmermann T, du Fay de Lavallaz J, Nestelberger T, Gualandro DM, Strebel I, Badertscher P, Lopez-Ayala P, Widmer V, Freese M, Miro O, Christ M, Cullen L, Than M, Martin-Sanchez FJ, Di Somma S, Peacock WF, Keller DI, Boeddinghaus J, Twerenbold R, Wussler D, Koechlin L, Walter JE, Burgler F, Geigy N, Kuhne M, Reichlin T, Lohrmann J, Mueller C. Incidence, characteristics, determinants, and prognostic impact of recurrent syncope. Europace. 2020 Dec 23;22(12):1885-1895. doi: 10.1093/europace/euaa227. PMID 33038231
- [Derived] Badertscher P, du Fay de Lavallaz J, Hammerer-Lercher A, Nestelberger T, Zimmermann T, Geiger M, Imahorn O, Miro O, Salgado E, Christ M, Cullen L, Than M, Martin-Sanchez FJ, Di Somma S, Peacock WF, Keller DI, Costabel JP, Walter J, Boeddinghaus J, Twerenbold R, Mendez A, Gospodinov B, Puelacher C, Wussler D, Koechlin L, Kawecki D, Geigy N, Strebel I, Lohrmann J, Kuhne M, Reichlin T, Mueller C; BASEL IX Investigators. Prevalence of Pulmonary Embolism in Patients With Syncope. J Am Coll Cardiol. 2019 Aug 13;74(6):744-754. doi: 10.1016/j.jacc.2019.06.020. PMID 31395124
- [Derived] du Fay de Lavallaz J, Badertscher P, Nestelberger T, Zimmermann T, Miro O, Salgado E, Christ M, Geigy N, Cullen L, Than M, Javier Martin-Sanchez F, Di Somma S, Frank Peacock W, Morawiec B, Walter J, Twerenbold R, Puelacher C, Wussler D, Boeddinghaus J, Koechlin L, Strebel I, Keller DI, Lohrmann J, Michou E, Kuhne M, Reichlin T, Mueller C; BASEL IX Investigators. B-Type Natriuretic Peptides and Cardiac Troponins for Diagnosis and Risk-Stratification of Syncope. Circulation. 2019 May 21;139(21):2403-2418. doi: 10.1161/CIRCULATIONAHA.118.038358. Epub 2019 Feb 25. PMID 30798615
- [Derived] du Fay de Lavallaz J, Badertscher P, Nestelberger T, Isenrich R, Miro O, Salgado E, Geigy N, Christ M, Cullen L, Than M, Martin-Sanchez FJ, Bustamante Mandrion J, Di Somma S, Peacock WF, Kawecki D, Boeddinghaus J, Twerenbold R, Puelacher C, Wussler D, Strebel I, Keller DI, Poepping I, Kuhne M, Mueller C, Reichlin T; BASEL IX Investigators; Gimenez MR, Walter J, Kozhuharov N, Shrestha S, Mueller D, Sazgary L, Morawiec B, Muzyk P, Nowalany-Kozielska E, Freese M, Stelzig C, Meissner K, Kulangara C, Hartmann B, Ferel I, Sabti Z, Greenslade J, Hawkins T, Rentsch K, von Eckardstein A, Buser A, Kloos W, Lohrmann J, Osswald S. Prospective validation of prognostic and diagnostic syncope scores in the emergency department. Int J Cardiol. 2018 Oct 15;269:114-121. doi: 10.1016/j.ijcard.2018.06.088. Epub 2018 Jun 21. PMID 30224031
- [Derived] Badertscher P, Nestelberger T, de Lavallaz JDF, Than M, Morawiec B, Kawecki D, Miro O, Lopez B, Martin-Sanchez FJ, Bustamante J, Geigy N, Christ M, Di Somma S, Peacock WF, Cullen L, Sarasin F, Flores D, Tschuck M, Boeddinghaus J, Twerenbold R, Wildi K, Sabti Z, Puelacher C, Rubini Gimenez M, Kozhuharov N, Shrestha S, Strebel I, Rentsch K, Keller DI, Poepping I, Buser A, Kloos W, Lohrmann J, Kuehne M, Osswald S, Reichlin T, Mueller C. Prohormones in the Early Diagnosis of Cardiac Syncope. J Am Heart Assoc. 2017 Dec 14;6(12):e006592. doi: 10.1161/JAHA.117.006592. PMID 29426039